CLINICAL TRIAL: NCT04993183
Title: Promoting an incLUsive Society Towards Older Adults With Physical Disabilities Through Disability Simulation Education (PLUS)
Brief Title: Promoting an incLUsive Society Towards Older Adults With Physical Disabilities
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Suzanne HS Lo, Assistant Professor, Chinese University of Hong Kong
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: PLUS
Record Dates: First submitted 2021-07-21; First posted 2021-08-06 (Actual); Last update posted 2024-04-15 (Actual); Status verified 2024-04

CONDITIONS: Disability Physical; Social Acceptance; Respect
Keywords: Physical disability; Social inclusion; Disability simulation; Education
MeSH Terms: conditions — Social Inclusion | interventions — Congresses as Topic

STUDY DESIGN:
Intervention Model Description: All recruited participants will receive the intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 3-day PLUS Convention (Experimental): Participants will participate in a 3-day PLUS Convention, comprising an inclusivity education workshop, service-learning seminar, disability simulation workshop, and two community contact sessions.
  Interventions: Behavioral: 3-day PLUS Convention

INTERVENTIONS:
Behavioral: 3-day PLUS Convention — Participants will participate in a 3-day PLUS Convention, comprising an inclusivity education workshop, a service-learning seminar, a disability simulation workshop, and two community contact sessions which will consist of a 60-minute interview with an older adult with a physical disability and an outdoor experience. Discussion sessions will be facilitated throughout to consolidate learning.

SUMMARY:
To improve secondary school students' positive attitudes towards older adults with physical disabilities via a Promoting an incLUsive Society towards older adults with physical disabilities through disability simulation education (PLUS) project.

DETAILED DESCRIPTION:
A pretest-posttest and qualitative study design will be adopted. 1,000 junior secondary students will be recruited from six secondary schools in Hong Kong by convenience sampling to participate in a 3-day PLUS Convention. Changes in students' attitudes towards older adults with physical disabilities and satisfaction with life, and their satisfaction with the disability simulation experience will be assessed. Semi-structured interviews will be conducted with students, facilitators, teachers, and older adults with physical disabilities to gain further feedback.

ELIGIBILITY:
Inclusion Criteria:

1. currently a secondary 1 to secondary 3 student
2. studying in a secondary school in Hong Kong
3. communicable in Cantonese
4. willing to attend all of the activities of the 3-day PLUS Convention

Exclusion Criteria:

1. have a physical or learning disability
2. diagnosed with a severe psychiatric illness

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 1111 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2024-03-31 (Actual)

PRIMARY OUTCOMES:
Change in the participants' attitudes towards older adults with physical disabilities | Change from baseline to immediately after completion of the intervention (2 months)
  The 47-item Students' Attitudes toward People with a Disability Scale will be used. It was developed locally in the Baseline Survey of Students' Attitudes towards People with a Disability, a study conducted by the Equal Opportunities Commission in Hong Kong. It encompasses four attitude sub-scales, namely social acceptance, behavioural misconceptions, pessimism-hopelessness, and optimism-human rights. Participants will rate their agreement with each item on a 4-point Likert scale (1 = "Strongly agree" - 4 = "Strongly disagree"). The four attitude sub-scale scores will then be converted along a scale between 1-100. A higher score will indicate a more positive attitude towards people with a disability. All sub-scales had Cronbach's Alpha scores ranging from 0.69 to 0.85, which support their respectable reliability.

SECONDARY OUTCOMES:
Change in the participants' level of life satisfaction | Change from baseline to immediately after completion of the intervention (2 months)
  The 5-item Satisfaction With Life Scale (SWLS) will be adopted. Participants will rate their overall judgement of their life on a 7-point Likert scale (1 = "Strongly disagree" - 7 = "Strongly agree"). The total score ranges from 5 to 35 points, with a higher score indicating a higher satisfaction with life. The SWLS has a Cronbach's Alpha score of 0.87, supporting its internal consistency and reliability.
The participants' level of satisfaction with the disability simulation workshop | Immediately after completion of the disability simulation workshop (within 1 day)
  The 18-item Satisfaction with Disability Simulation Experience Scale (SDSES) will be used. Participants will rate their extent of agreement with the simulations using a 5-point Likert scale (1 = "Strongly disagree" - 5 = "Strongly agree") to indicate their satisfaction with them. A higher score will indicate higher satisfaction with the simulation experience. The survey will have one open-ended question asking students to provide additional comments about their simulation experience. The scale's internal consistency reliability is supported as its whole Cronbach's coefficient values ranged from 0.70 to 0.88.

CONTACTS AND LOCATIONS:
Overall Officials: Suzanne Lo, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Secondary Schools, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Yes
The datasets used and/or analysed during the current study will be available from the corresponding author on reasonable request.
Supporting Information: Study Protocol, ICF
Time Frame: The datasets used and/or analysed during the current study will be available from the corresponding author, on reasonable request, for six years upon completion of the study
Access Criteria: The datasets used and/or analysed during the current study will be available from the corresponding author on reasonable request.